CLINICAL TRIAL: NCT05151796
Title: Effect of Continuation of Aspirin Before Isolated Heart Valve Surgery on Postoperative Bleeding and Transfusion: a Single-center Retrospective Study
Brief Title: Continuation of Aspirin Before Isolated Heart Valve Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor of Anesthesia, University of Liege
Other Study IDs: ulganescardio_aspirine
Record Dates: First submitted 2021-10-05; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Isolated Heart Valve Surgery
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspirin continued within 5 days before surgery
  Interventions: Drug: Aspirin
- Aspirin discontinued more than 5 days before surgery

INTERVENTIONS:
Drug: Aspirin — Daily aspirin intake for cardiovascular prevention
  Groups: Aspirin continued within 5 days before surgery

SUMMARY:
Whether or not continuing aspirin up to de day before surgery increases the risk of bleeding and/or prevents thrombo-embolic complications remains debated. The investigators retrospectively investigated the whether continuing aspirine within 5 days of isolated heart valve surgery increased the risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Isolated heart valve surgery

Exclusion Criteria:

* Antiplatelet agent other than aspirin or anticoagulant not discontinued preoperatively
* Emergent or salvage surgery
* Surgery for endocarditis
* Use of NSAIDs within 48 hours before surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing isolated heart valve surgery at the University Hospital of Liege (Belgium)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of units of packed red blood cells transfused anytime during the hospital stay | 30 days

SECONDARY OUTCOMES:
Chest tube drainage | 24 hours
  volume of chest tube drainage
Surgical revision for bleeding | 24 hours
Any thrombo-embolic complication | 30 days
Transfusion of any type of blood product | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bonhomme, MD, PhD, Study Chair — CHU of Liège
Locations (1):
- CHU of Liege, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houben AM, Crepy M, Senard M, Bonhomme V, Tchana-Sato V, Hans G. Preoperative continuation of aspirin before isolated heart valve surgery and postoperative bleeding and transfusion: a single-center retrospective study. Acta Chir Belg. 2024 Aug;124(4):274-280. doi: 10.1080/00015458.2023.2298097. Epub 2023 Dec 26. PMID 38146908